CLINICAL TRIAL: NCT02575157
Title: Changes in Biochemical Markers of Bone Turnover (Serum CTX and PlNP) After Initiation of a "Drug Holiday" From Bisphosphonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Bone Health Alliance (Other)
Collaborators: Roche Pharma AG (Industry); National Osteoporosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: NBHADH1
Record Dates: First submitted 2015-10-10; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Discontinuing usage (No Intervention): Patients will discontinue use of bisphosphonates. Bone markers and BMD will be monitored until a need for reinitiation of treatment within 2-years is identified or needed.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Bisphosphonates (BP) are widely used in the prevention and treatment of osteoporosis in postmenopausal women and older men. Recently, there has been concern about the risk of adverse events after several years of using these agents. This has resulted in a publication from the Food and Drug Administration that suggested that, for many individuals, a holiday from bisphosphonates might be considered after 4-5 years of continuous use. In that publication there was little, if any, guidance on how clinicians should proceed after the holiday is initiated.

DETAILED DESCRIPTION:
Bisphosphonates (BP) are widely used in the prevention and treatment of osteoporosis in postmenopausal women and older men. Recently, there has been concern about the risk of adverse events after several years of using these agents. This has resulted in a publication from the Food and Drug Administration that suggested that, for many individuals, a holiday from bisphosphonates might be considered after 4-5 years of continuous use. In that publication there was little, if any, guidance on how clinicians should proceed after the holiday is initiated.

Bisphosphonates likely work by first binding to the hydroxyapatite crystal, and when the crystal is dissolved in the acid medium created by osteoclasts in the process of bone resorption, the bisphosphonate is released, and is incorporated into the osteoclast where it inhibits farnesyl pyrophosphate synthase and interferes with intracellular protein trafficking. The consequence is loss of osteoclast resorptive activity and in some cases osteoclast apoptosis. Thus the potency of any particular bisphosphonate is dependent on independent processes, such as the binding affinity to hydroxyapatite and the potency of enzyme inhibition. As patients remain on bisphosphonates, it is likely that more and more of the drug will become incorporated into the skeleton. Therefore, when the drugs are discontinued, they gradually leach from the skeleton. The rate at which the effects of the drug wear off ("off-rate"), as evidenced by changes in biochemical markers of bone turnover, should be dependent on the binding affinity. The length of time for which the pharmacologic effect continues will also be dependent on potency of enzyme inhibition. Thus, each bisphosphonate will likely have a unique off-rate. Data from the extensions of some of the clinical trials support the concept of variable off rates, but there are no head to head data to determine this. Furthermore, clinical trial data may have limited utility in patients seen in a practice setting.

Biochemical markers have been shown in a number of studies to be reliable surrogate markers for the overall rate of bone remodeling in the skeleton. After menopause or ovariectomy, serum levels of biochemical markers increase and these increments have been associated with the rate of bone loss as measured by dual x-ray absorptiometry (DXA). As individuals age, fracture risk is determined by both age and bone mineral density (BMD). Trabecular bone score (TBS), an advanced application for DXA, describes the quality of bone microarchitecture, which has been shown to impact bone strength and thus fracture risk.

In clinical trial data where bisphosphonates have been discontinued and subjects continue to be followed, biochemical markers increase after the drug is stopped, and presumably the fracture benefit of the drug will be gradually lost. Concern over possible association of the long term side effects of bisphosphonates (notably osteonecrosis of the jaw and atypical fractures of the femoral shaft) have led to a concept, endorsed by FDA, of a drug holiday. At present there are no guidelines on how patients should be followed when the drugs are discontinued. From the clinical trial data in different subject populations with differing protocols, as well as in vitro data, the inference may be drawn that the off effects will vary with different drugs. It is hypothesized that risedronate will lose its effect more rapidly than alendronate. However, this concept has never been studied in a prospective clinical study. Therefore, the intent in this prospective study is to examine patients who are about to be taken off of 2 different bisphosphonate drugs and compare their off rates using two established biochemical markers (sCTX and P1NP).

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women or males >50 years who have taken oral bisphosphonates (risedronate or alendronate) for five years or more, and in whom it is considered reasonable to initiate a holiday from the medication, or those who have been on a holiday for up to 3 months will be eligible for screening visit.
2. Subjects whose 25(0H) D level is above 30 ng/ml (subjects with 25(0H)D from 10-29 ng/ml may be included after supplementation and assessment of serum 25(0H)D) level is above 30 ng/ml.

   -

Exclusion Criteria:

1. Current steroid treatment at or greater than 5 mg/day prednisone or equivalent.
2. The use of any other bone active medication other than risedronate or alendronate.
3. The use of teriparatide within the past 4 years.
4. A contra-indication to the discontinuation of bisphosphonate (e.g. fracture during treatment, extremely low t-score).
5. Subjects with fasting serum sCTX less than 100 pg/ml or greater than 300 pg/mL while taking bisphosphonates.
6. Failure to bring 25(0H)D serum level to 30 ng/ml or greater.
7. Metabolic bone disease other than osteoporosis.
8. Abnormal thyroid function (may be included when thyroid function is shown to be normal by TSH). Per local lab assessment.
9. Evidence of failure to adhere to bisphosphonate use -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Changes in bone turnover markers. | 2 years
Changes in bone mineral density | 2 years
Changes in trabecular bone score | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Taylor C. Wallace, Washington D.C., District of Columbia, United States